CLINICAL TRIAL: NCT02633930
Title: Helicobacter Pylori Eradication With Berberine Hydrochloride, Lansoprazole, Amoxicillin and Bismuth Versus Clarithromycin Bismuth, Lansoprazole and Amoxicillin: A Randomized, Open-label, Non-inferiority, Phase Ⅳ Trial
Brief Title: Helicobacter Pylori Eradication With Berberine Quadruple Therapy Versus Clarithromycin Quadruple Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Doctor of Xijing Hospital of Digestive Diseases,Principal investagator,Clinical professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20151203-2
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Gastritis; Peptic Ulcer; Dyspepsia
Keywords: helicobacter pylori; berberine-containing quadruple therapy; clarithromycin-containing quadruple therapy
MeSH Terms: conditions — Gastritis; Peptic Ulcer; Dyspepsia | interventions — Berberine; Clarithromycin; Bismuth; Lansoprazole; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- berberine quadruple therapy (Experimental): Berberine 300 mg, three times daily for 14 days,lansoprazole 30 mg,amoxicillin 1000 mg, and Bismuth 220 mg by mouth, twice daily for 14 days.
  Interventions: Drug: Berberine; Drug: Bismuth; Drug: Lansoprazole; Drug: amoxicillin
- clarithromycin quadruple therapy (Active Comparator): Bismuth 220 mg, lansoprazole30 mg, amoxicillin 1000 mg, and clarithromycin 500 mg by mouth,twice daily for 14 days.
  Interventions: Drug: clarithromycin; Drug: Bismuth; Drug: Lansoprazole; Drug: amoxicillin

INTERVENTIONS:
Drug: Berberine — : given for 14 days at a dose of berberine 100 mg 3 tablets TID, lansoprazole 30 mg BID, amoxicillin 500 mg 2 capsules BID, and colloidal bismuth tartrate capsule55 mg 4 capsules BID
  Arms: berberine quadruple therapy
Drug: clarithromycin — Clarithromycin-containing quadruple therapy group 500 mg 1 tablet BID plus amoxicillin 500 mg 2 capsules BID, lansoprazole 30mg 1tablet BID, and colloidal bismuth tartrate capsule55 mg 4 capsules BID.
  Arms: clarithromycin quadruple therapy
Drug: Bismuth — Bismuth:given for 14 days at a dose of colloidal bismuth tartrate capsule 55 mg 4 capsules BID, lansoprazole30 mg BID, amoxicillin 500 mg 2 capsules BID, and clarithromycin 500 mg 1 tablet BID or given for 14 days at a dose of colloidal bismuth tartrate capsule 55 mg 4 capsules BID, lansoprazole30 mg BID, amoxicillin 500 mg 2 capsules BID, and berberine 100 mg 3 tablet TID
  Other Names: Bitnal
Drug: Lansoprazole — Lansoprazole 30mg 1tablet BID plus amoxicillin 500 mg 2 capsules BID, clarithromycin 500 mg 1 tablet BID, and colloidal bismuth tartrate capsule 55 mg 4 capsules BID or berberine 100 mg 3 tablets TID given to berberine-containing quadruple therapy group or clarithromycin-containing quadruple therapy group
  Other Names: Takepron
Drug: amoxicillin — Amoxicillin 500 mg 2 capsules BID plus lansoprazole 30mg 1tablet BID, clarithromycin 500 mg 1 tablet BID, and colloidal bismuth tartrate capsule 55 mg 4 capsules BID or berberine 100 mg 3 tablets TID as a dose given for clarithromycin-containing quadruple therapy or berberine-containing quadruple therapy.
  Other Names: Amoxy ( Uni-Amocin )

SUMMARY:
This study aims at evaluating efficacy and safety of berberine-containing quadruple therapy(berberine, lansoprazole, bismuth and amoxicillin) versus clarithromycin-containing quadruple therapy (clarithromycin,lansoprazole, bismuth and amoxicillin) in H. pylori eradication. It is hypothesized that berberine-containing quadruple therapy is non-inferior to clarithromycin-containing quadruple therapy. Patients with confirmed H. pylori positive status will be randomized to one of the treatments described above. At week 2 and 6 follow-up visits, a urea breath test(UBT) will be performed to confirm eradication.

DETAILED DESCRIPTION:
The study will include three phases: screening, treatment and follow-up. Screening: this phase will last a maximum of 28 days and subjects eligibility will be evaluated after informed consent signature. Endoscopy and Urea Breath test will be performed in addition to the baseline routine evaluations.

Treatment: Subjects are randomly assigned to treatment and will be treated for 14 days. A randomization visit will take place on Day 0 and an end-of-treatment visit will take place between day 12 and 14.

Follow-up: includes two visits. approximately 14 days of treatment and 28 days after the end of treatment. Eradication of H. Pylori will be confirmed through urea breath test(UBT).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18~70,both gender.
2. Patients with upper gastrointestinal symptoms and with documented H.pylori infection.
3. Patients are willing to receive eradication treatment.
4. Women are eligible if they are not pregnant or nursing, and if they are of childbearing potential they are required to use medically acceptable contraception for the duration of the study and 30 days thereafter.

Exclusion Criteria:

1. Patients are excluded if they have previously used antibiotics to eradicate adequately recorded infection with H. pylori.
2. Contraindications to study drugs.
3. Substantial organ impairment, severe or unstable cardiopulmonary or endocrine disease.
4. Constant use of anti-ulcer drugs ( including taking proton-pump. inhibitors(PPI) within 2 weeks before the [13C] urea breath test), antibiotics or bismuth complexes (more than 3 times /1 month before screening)
5. Pregnant or lactating women.
6. Underwent upper gastrointestinal Surgery.
7. Patients with Barrett esophageal or highly atypical hyperplasia, have symptom of dysphagia.
8. Evidence of bleeding or iron efficiency anemia.
9. A history of malignancy.
10. Drug or alcohol abuse history in the past 1 year.
11. Systemic use of corticosteroids, non steroidal anti-inflammatory drugs, anticoagulants, platelet aggregation inhibitors (except the use of aspirin for less than 100 mg/d).
12. Enrolled in other clinical trials in the past 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
helicobacter pylori eradication | 28 days after treatment
  The primary end point of this study is H.pylori eradication,established by negative [13C] urea breath test 28 days after the end of eradication.

SECONDARY OUTCOMES:
symptoms effective rates | 14 days of treatment, and 28 days after treatment
  Evaluation effective rate of symptoms 2 weeks of treatment and 4 weeks after the end of treatment.
  Symptom effective rate =（total score before treatment - total score after treatment）/total score before treatment x 100%. Total score = frequency + severity.
  Frequency score is calculated by all the frequency of heartburn, reflux, abdominal pain, and flatulence. Severity is accumulated by the degree of symptoms described above, which is divided to 4 degree as 0 presenting none, and 3 presenting most severe
adverse events | 14 days of treatment, and 28 days after treatment
  Participants with Adverse Events as a Measure of Safety and Tolerability.The common side effects of the study include headache, dizziness, skin rash, other gastrointestinal disorders, pyrexia, cough and back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Shi, Ph. D, Principal Investigator — Xijing Hospital
Locations (2):
- China (2):
  - Xijing Hospital of Digestive Diseases, Xi’an, Shanxi
  - Xijing Hospital of Digestive Disease, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No